CLINICAL TRIAL: NCT00003716
Title: Phase II Trial of Rituximab in Patients With B-Cell Lymphoproliferative Disorders Associated With Pharmacologic Immunosuppression
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Lymphoproliferative Disorder Associated With Immunosuppression Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066825; SUMC-03; NCI-V98-1508
Record Dates: First submitted 1999-11-01; First posted 2003-12-05 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma
Keywords: childhood Burkitt lymphoma; childhood immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab in treating patients who have lymphoproliferative disorder that is associated with immunosuppression therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of rituximab in patients with B-cell lymphoproliferative disorders while under pharmacologic immune suppression for control of either allograft rejection or autoimmune disease. II. Evaluate the safety and direct toxicity of rituximab in this patient population, including the potential for opportunistic infections. III. Evaluate the secondary consequences of rituximab therapy in this population, including changes in the requirement for immunosuppressive drugs, effects on graft rejection, graft survival, and severity of autoimmune disease.

OUTLINE: Patients receive rituximab IV over several hours. Treatment repeats every week for 4 courses. Patients are followed every month for 6 months, and then every 3 months until relapse or 2 years.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Polyclonal or monoclonal B-cell lymphoproliferative disorder while under pharmacologic immune suppression for control of either allograft rejection or autoimmune disease Measurable disease as defined by one of the following: At least 1 tumor mass measuring 1.0 cm in largest dimension Greater than 25% marrow involvement Quantifiable extranodal disease Expression of CD20 antigen confirmed by biopsy or fine needle aspirate Progression of disease or stable disease following reduction of immunosuppressive medication and antiviral therapy Inability to further reduce immunosuppressive medication

PATIENT CHARACTERISTICS: Age: 3 to 70 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hepatic: Not specified Renal: Not specified Cardiovascular: No congestive heart failure Pulmonary: No pneumonitis Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No serious nonmalignant disease No active uncontrolled bacterial, viral, or fungal infections

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) No concurrent chemotherapy Endocrine therapy: At least 2 weeks since change in dosing and type of immunosuppressive drugs unless due to progression of disease Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery (except diagnostic surgery) Other: At least 30 days or 5 half-lives since other prior investigational drugs or whichever is longer

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-03 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States